CLINICAL TRIAL: NCT05005377
Title: Peri-Implant Soft and Hard Tissue Stability After Loading of Implants Following Socket Preservation With Platelet-Rich Fibrin and Freeze-Dried Bone Allograft
Brief Title: Peri-Implant Soft and Hard Tissue Stability Following Socket Preservation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1396.261
Record Dates: First submitted 2021-07-15; First posted 2021-08-13 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-07

CONDITIONS: Alveolar Ridge Augmentation; Bone Transplantation

STUDY DESIGN:
Intervention Model Description: 48 patients were randomly divided into two groups for anterior ridge preservation with PRF and FDBA. At 12 months after implant placement and prosthetic delivery, bone loss was evaluated radiographically while soft tissue changes were evaluated by measuring gingival recession, papilla index, and bleeding on probing (BOP).
Who Masked: Investigator
Masking Description: The investigator who analyzed the data was blinded from the procedure ( The participants were assigned to A and B groups and it was not clear for the investigator which data belonged to which procedure).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Socket Preservation with Platelet-Rich Fibrin (Experimental): 10cc of blood was drawn from each patient and centrifuged at 2700 revolutions per minute (rpm) for 12 minutes to obtain PRF. The extraction socket was filled with PRF and covered using a membrane made of PRF.
  Interventions: Procedure: Socket Preservation with Platelet-Rich Fibrin
- Socket Preservation with Freeze-Dried Bone Allograft (Experimental): the extraction socket was filled with FDBA (CenoBone®; Tissue Regeneration Corp., Kish Island, Iran) without flap elevation. The socket was covered using a free palatal mucosal graft obtained by the pouch technique.
  Interventions: Procedure: Socket Preservation with Freeze-Dried Bone Allograft

INTERVENTIONS:
Procedure: Socket Preservation with Platelet-Rich Fibrin — 10cc of blood was drawn from each patient and centrifuged at 2700 revolutions per minute (rpm) for 12 minutes to obtain PRF. The extraction socket was filled with PRF and covered using a membrane made of PRF.
  Arms: Socket Preservation with Platelet-Rich Fibrin
Procedure: Socket Preservation with Freeze-Dried Bone Allograft — The extraction socket was filled with FDBA (CenoBone®; Tissue Regeneration Corp., Kish Island, Iran) without flap elevation. The socket was covered using a free palatal mucosal graft obtained by the pouch technique.
  Arms: Socket Preservation with Freeze-Dried Bone Allograft

SUMMARY:
The viability of Platelet Rich Fibrin (PRF) on enhancement of osseous and associated tissue healing has been substantiated well in literature. This study aimed to assess peri-implant soft and hard tissue changes after prosthetic loading of implants following socket preservation with platelet-rich fibrin (PRF) and freeze-dried bone allograft (FDBA) in a 12-month period.

This Study evaluated 48 patients who were randomly divided into two groups for anterior ridge preservation with PRF and FDBA. At 12 months after implant placement and prosthetic delivery, bone loss was evaluated radiographically while soft tissue changes were evaluated by measuring gingival recession, papilla index, and bleeding on probing (BOP). The differences between the PRF and FDBA groups were analyzed using Fisher's exact test and student's t-test (P<0.05).

DETAILED DESCRIPTION:
This study was conducted on 48 patients over 18 years of age (average age of 38 years). The patients required single-rooted incisor/premolar teeth extraction with a hopeless prognosis; for whom, socket preservation with PRF or FDBA was later performed. The reasons for tooth extraction included root fracture, failed root canal therapy, and extensive non-restorable caries. The ethics and study design was approved the Research Ethics Committee of Tehran University of Medical Sciences (IR.TUMS.DENTISTRY.REC.1396.2610) and conducted in accordance with the Declaration of Helsinki. All patients signed an informed consent prior to enrollment. They were free to leave the study at any time and ensured about the confidentiality of their information. The exclusion criteria included a history of systemic disease and head/neck radiotherapy, use of drugs affecting bone metabolism, smoking more than 10 cigarettes per day, the presence of significant periapical or periodontal lesions around the respective teeth, and the presence of dehiscence or fenestration larger than 3mm in the buccal bone plate. After extraction of the teeth, the patients underwent socket preservation with the use of PRF or FDBA. 4 months later, they received a Zimmer ScrewVent bone-level implant (Zimmer, Biomet, USA) which was left in place for 2 to 4 month (mandible and maxilla respectively) to achieve proper osseointegration. All implants were successfully osseointegrated. 10 patients were excluded during the study due to poor cooperation in the follow-up period. Eventually, 38 patients including 23 females and 15 males were subjected to hard and soft tissue assessments at 6 and 12 months, postoperatively. Patients in the PRF group included 9 males and 9 females (a total of 18) with a mean age of 30.81 years (ranging from 21 to 50 years). Patients in the FDBA group included 6 males and 14 females (a total of 20) with a mean age of 37.25 years (ranging from 22 to 50 years).

In second-stage surgery, a full-thickness flap was elevated and a gingival former (Zimmer, Biomet, USA) matching the fixture size placed. Soft tissue healing around the gingival former was allowed for 3 weeks and then a fixture level impression made using the closed-tray impression technique by additional silicone (Panasil, Kettenbach GmbH & Co. KG, Eschenburg). The master cast was poured with G-mask SnowRock (Velmix; MungyoGroup, Korea) and Moldano dental stone (Tara, Iran). All selected abutments were straight, with a 0.5 mm gingival height. If the gingival height around an implant was variable, the higher value was chosen and other surfaces of the abutment were prepared such that the final finish line was positioned 0.5 mm subgingivally. After abutment preparation, a metal framework was waxed-up for a cement-retained metal-ceramic crown using resin pattern (GC Corporation, USA). The framework was then cast (Wirobond® C, Bego, USA) and tried in the second session. Vita Classic Shade Guide (Vitapan, Germany) was used to select the tooth shade. Porcelain adjustments (VITA VM ceramic, VITA Zahnfabrik, Germany) including the contacts, occlusion, contour and the esthetic appearance of the crown was performed at the third session. The crowns were then glazed. In the fourth prosthetic session, the abutments were tighten to 25 N.Cm final torque and sealed with a Teflon band. The glazed crown was cemented with temporary cement (TempBond, Kerr) and excess cement thoroughly removed. Complete seating of the crown and excess cement removal were ensured in the first radiograph.

To assess the hard tissue stability around each implant, a digital radiograph (Digora Optime, Acteon, India) was obtained with a size 2 sensor using a film holder (Kerr). All baseline and follow-up radiographs were parallel and exposure settings were the same for each patient in the baseline and follow-up radiographs. Using Scanora software (SCANORA lite, Soredex, Helsinki, Finland), the distance from the crestal bone-fixture interface to the abutment-crown interface (crown margin) was measured at the mesial and distal surfaces of the implant at 0, 6 and 12 months after implant placement (Fig1).These measurements were repeated 3 times at the mesial and 3 times at the distal surfaces for each patient and the mean values reported to minimize the errors. To assess soft tissue changes, clinical gingival parameters including the gingival recession (defined as the change in the distance from the gingival margin to the crown margin compared with time 0), the papilla index (distance from the tip of the papilla to the crown margin in the mesial and distal surfaces) (Fig2), and bleeding on probing (BOP) at the mesiobuccal and distobuccal points were measured at 0, 6 and 12 months, postoperatively.

Data were analyzed using SPSS version 22. Qualitative variables were compared using Fisher's exact test while quantitative variables were compared using unpaired student's t-test. The level of significance was set at 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age, who were referred for extraction of the hopeless teeth. The reasons for tooth extraction included root fracture, failed root canal therapy, and extensive non-restorable caries.

Exclusion Criteria:

* a history of systemic disease and head/neck radiotherapy, use of drugs affecting bone metabolism, smoking more than 10 cigarettes per day, the presence of significant periapical or periodontal lesions around the respective teeth, and the presence of dehiscence or fenestration larger than 3mm in the buccal bone plate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
mean vertical ridge resorption | 0 month
  Mean bone loss around implants measured using Scanora software (SCANORA lite, Soredex, Helsinki, Finland), the distance from the crestal bone-fixture interface to the abutment-crown interface (crown margin) was measured at the mesial and distal surfaces of the implant immediately after implant placement. These measurements were repeated 3 times at the mesial and 3 times at the distal surfaces for each patient and the mean values reported to minimize the errors.
mean vertical ridge resorption | 6 month
  Mean bone loss around implants measured using Scanora software (SCANORA lite, Soredex, Helsinki, Finland), the distance from the crestal bone-fixture interface to the abutment-crown interface (crown margin) was measured at the mesial and distal surfaces of the implant 6 months after implant placement. These measurements were repeated 3 times at the mesial and 3 times at the distal surfaces for each patient and the mean values reported to minimize the errors.
mean vertical ridge resorption | 12 month
  Mean bone loss around implants measured using Scanora software (SCANORA lite, Soredex, Helsinki, Finland), the distance from the crestal bone-fixture interface to the abutment-crown interface (crown margin) was measured at the mesial and distal surfaces of the implant 12 months after implant placement. These measurements were repeated 3 times at the mesial and 3 times at the distal surfaces for each patient and the mean values reported to minimize the errors.
Mean Gingival Recession | 0 month
  gingival recession was defined as the changes in the distance from the gingival margin to the crown margin )
Mean Gingival Recession | 6 month
  gingival recession was defined as the changes in the distance from the gingival margin to the crown margin compared with time 0)
Mean Gingival Recession | 12 month
  gingival recession was defined as the changes in the distance from the gingival margin to the crown margin compared with time 0)
Changes in Papilla Index | 0 month
  it was measured via the distance from the tip of the papilla to the crown margin in the mesial and distal surfaces of the restoration
Changes in Papilla Index | 6 month
  it was measured via the distance from the tip of the papilla to the crown margin in the mesial and distal surfaces of the restoration
Changes in Papilla Index | 12 month
  it was measured via the distance from the tip of the papilla to the crown margin in the mesial and distal surfaces of the restoration
Frequency of bleeding on probing | 0 month
  was measured at the mesiobuccal and distobuccal points of the restoration
Frequency of bleeding on probing | 6 month
  was measured at the mesiobuccal and distobuccal points of the restoration
Frequency of bleeding on probing | 12 month
  was measured at the mesiobuccal and distobuccal points of the restoration

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Azangookhiavi H, Habibzadeh S, Zahmatkesh H, Mellati E, Mosaddad SA, Dadpour Y. The effect of platelet-rich fibrin (PRF) versus freeze-dried bone allograft (FDBA) used in alveolar ridge preservation on the peri-implant soft and hard tissues: a randomized clinical trial. BMC Oral Health. 2024 Jun 14;24(1):693. doi: 10.1186/s12903-024-04478-1. PMID 38877446